CLINICAL TRIAL: NCT01153750
Title: Phase II Study to Evaluate the Efficacy of a Chemotherapy Combination With Imatinib (Glivec®) and 5-FU/Leucovorin in Patients With Advanced Carcinoma of the Gallbladder and Bile Duct
Brief Title: Efficacy of Imatinib and 5-FU/Leucovorin in Patients With Advanced Carcinoma of the Gallbladder and Bile Duct
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Dresden (Other)
Responsible Party: PD Dr. Jan Stoehlmacher, University Hospital Dresden, Medical Department I
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-Glivec-012
Record Dates: First submitted 2010-04-01; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-04

CONDITIONS: Advanced or Metastatic Cholangiocellular Carcinoma and Bile Duct
Keywords: cholangiocellular carcinoma; bile duct cancer
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glivec and 5-Fluorouracil/Leucovorin (Experimental): All patients will receive Glivec® 600 mg once daily without dose escalation. Glivec® will be given on day -4, -3, -2, -1, 1, 2, 3 and 4. There will be no day "0". Patients will also receive 5-FU (2000mg/qm 24hc.i. d1 + d2) and leucovorin (200mg/qm 2h-infusion) qd15.
  Interventions: Drug: Glivec

INTERVENTIONS:
Drug: Glivec

SUMMARY:
To test the efficacy of a combination chemotherapy of imatinib and 5-FU in advanced or metastatic cholangiocellular carcinoma.

DETAILED DESCRIPTION:
Efficacy: Tumor assessments should be performed by a CT or MRI scan, throughout the study. All assessments should be performed within 14 days of the scheduled day according to the visit schedules, and whenever clinically indicated otherwise. Radiological studies must use the same techniques as used at baseline. Evaluation will be based on RECIST criteria.

Safety: Safety assessments will consist of evaluating adverse events and serious adverse events, laboratory parameters including hematology, chemistry, vital signs, physical examinations, and documentation of all concomitant medications and/or therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/Cytologically confirmed diagnosis of advanced / metastatic carcinoma of the gallbladder or bile duct, which is unresectable or metastatic and therefore incurable with any conventional multimodality approach
* Performance status 0, 1 or 2 (ECOG)
* Written, voluntary informed consent
* Age > 18 years
* Adequate bone marrow function (Granulocytes > 1,5 x 109/l, Hb > 10 g/dl, Platelets > 100 x 109/l)
* Adequate hepatic and renal function ( bilirubin < 1,25 x upper normal limit or < 1,5 x upper normal limit if hyperbilirubinemia is related to underlying disease, ALAT + ASAT < 1,5 x upper normal limit, in case of liver metastases < 5 x upper normal limit, creatinine < 1,25 x upper normal limit)
* Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Female patients with child-bearing potential must perform a highly effective barrier method of birth control throughout the study with a proven efficacy of >99%. The contraception treatment should be performed for an additional six month following discontinuation from study treatment. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following discontinuation of study drug.

Exclusion Criteria:

* Patient has received any other investigational agents within 28 days of first day of study drug dosing.
* Patient is < 5 years free of another primary malignancy, except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ.
* Female patients who are pregnant or breast-feeding.
* Patient has a severe and/or uncontrolled medical disease.
* The concurrent use of warfarin or acetaminophen are not allowed with imatinib mesylate and need to be replaced by other medications (e.g. by low molecular heparins in case of warfarin).
* Radiotherapy or any major abdominal or thoracic surgery < 4 weeks before study entry (excluding diagnostic biopsy or port implantation)
* Patient has received neoadjuvant imatinib mesylate or fluoropyrimidines prior to study entry
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
* Known incompatibility of imatinib,5-FU, or leucovorin
* Known brain metastases
* Concurrent systemic chemotherapy, immunotherapy, hormone therapy
* History of severe psychiatric illness
* Drug- or alcohol abuse
* Patient has know chronic liver disease (i.e., chronic active hepatitis, and cirrhosis)
* Patients with dihydropyrimidine dehydrogenase deficiency (i.e. Treatment with Zostex)
* Patients that are associated with or dependent of the investigator or sponsor
* Patients with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
* Patients with a creatinine clearance of < 50ml/min.
* Patients with a severe decrease of bone marrow function
* Patients with acute infections
* Patients with severe decrease of liver function
* Patients in reduced performance status (ECOG > 2)
* No active vaccinations should be performed while being on study treatment
* Anemia caused by vitamin B12 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR)

SECONDARY OUTCOMES:
Progression-free survival (PFS)
Response rate (RR)
Overall survival
Toxicity
Evaluation of molecular predictive markers for response and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stoehlmacher, PD Dr., Principal Investigator — University Hospital Dresden
Locations (8):
- Germany (8):
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - University Hospital, Dresden, Saxony
  - University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Onkologische Schwerpunktpraxis Eppendorf, Hamburg
  - Staedtisches Klinikum Magdeburg, Magdeburg
  - Johannes-Gutenberg-Universität Mainz, Medical Department I, Mainz
  - Ruppiner Kliniken GmbH, Neuruppin
  - Praxisgemeinschaft Dr. Hancken und Partner, Stade